CLINICAL TRIAL: NCT04397471
Title: A Study to Collect Bone Marrow for Process Development and Production of Bone Marrow Mesenchymal Stromal Cells to Treat Severe COVID19 Pneumonitis
Brief Title: A Study to Collect Bone Marrow for Process Development and Production of BM-MSC to Treat Severe COVID19 Pneumonitis
Acronym: COMET20d
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: CCTU- Cancer Theme (Other)
Collaborators: Cambridge Cellular Therapies Laboratory (Unknown); The Evelyn Trust (Unknown)
Responsible Party: Sponsor-Investigator, CCTU- Cancer Theme, Dr Andrew McCaskie, Cambridge University Hospitals NHS Foundation Trust
Organization: Cambridge University Hospitals NHS Foundation Trust (Other)
Other Study IDs: COMET20d
Record Dates: First submitted 2020-05-13; First posted 2020-05-21 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Healthy Volunteers for Bone Marrow Donation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bone Marrow harvested from healthy donor volunteers to develop and manufacture cell-based therapy for COVID-19 pneumonitis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Volunteer: A one time only 30-80 mL sample of bone marrow will be collected from both posterior superior iliac crests.
  Interventions: Procedure: Bone Marrow Harvest

INTERVENTIONS:
Procedure: Bone Marrow Harvest — Healthy volunteer bone marrow harvest

SUMMARY:
The COVID-19 pandemic, commonly referred to as "coronavirus", first began in the city of Wuhan, China in December 2019. This virus has since spread globally, with infections reported in nearly every country. COVID-19 targets the body's respiratory system, where infections can be found in the nose, throat and lungs. The effect of COVID-19 infection is very variable, where many people might not know that they have been infected and have recovered from COVID-19. However, COVID-19 infection can cause people to have difficulty breathing. This can be severe enough to require hospitalisation and potentially intensive care treatment.

While they are being treated in hospital, COVID-19 infected patients can be found to have inflamed tissue in their lungs (referred to medically as "pneumonitis"). This inflammation is thought to be caused by their body's immune systems overacting to the infection rather than the COVID-19 virus itself. By potentially dampening down this overreaction of their immune system, it is hoped that COVID-19 patients with inflamed lungs have better and quicker chance to survive.

Mesenchymal stromal cells (MSCs) have been shown to have anti-inflammatory and healing properties on injured tissue. MSCs have been trialled in various diseases but have not yet been tested on patients with COVID-19. In this study, the investigators will obtain bone marrow from healthy volunteers to develop a cell-based treatment for COVID-19-related pneumonitis. The investigators will also determine whether it is feasible to recruit bone marrow donors in a clinically useful timeframe to treat COVID-19 patients. A future trial, COMET20, will use the bone marrow-derived MSCs (BM-MSCs) manufactured in COMET20d to treat COVID-19 patients suffering with pneumonitis, to determine whether the BMMSCs can reduce the likelihood for mechanical ventilation and reduce hospitalisation.

ELIGIBILITY:
Inclusion Criteria:

* Have given written informed consent to participate
* Be aged between 18 and 40 years old
* Have Eastern Cooperative Oncology Group (ECOG) performance status 0
* Be negative for mandatory infectious disease markers (IDM) as per World Marrow Donor Association (WMDA) guidelines
* Present a negative SARS-CoV2 screen
* Show absence of clinical symptoms of COVID-19 (Not have been in known COVID-19 contact within the previous 14 days, Adherence to national social distancing guidelines for 14 days)
* Have a BMI <35kg/m^2
* Women of childbearing potential need a negative pregnancy test (urine or blood) within 7 days prior to the marrow collection

Exclusion Criteria:

* Any major disease which would represent a contraindication to bone marrow donation based on WMDA guidelines
* Presence of any previous or active malignancy (other than non-melanoma skin cancer)
* Any other concurrent severe and/or uncontrolled medical condition
* Women who are pregnant or breast-feeding
* Any acute or chronic back complaint
* Presence of anaesthetic risk factors

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy adults aged 18-40 years who are negative for mandatory infectious disease markers including current COVID-19 infection.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2020-05 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Determine feasibility of recruiting healthy volunteers in a clinically useful timeframe. | 3 or more participants recruited in 1 month
  Successful identification of healthy volunteers in acceptable timeframe (i.e. within days) to donate bone marrow.
Manufacture a cell-based product suitable for clinical use | Successfully opening the next phase of the trial in approx. 2 months
  Successful manufacture of bone marrow-mesenchymal stromal cells suitable for clinical use

SECONDARY OUTCOMES:
Establishment of a robust process of production | Successfully opening the next phase of the trial in approx. 2 months
  Ability to prepare a dossier acceptable to the MHRA. Success will achieved if the dossier is deemed acceptable.
Production of stability data to be used in the MHRA dossier for the COMET clinical trial. | Successfully opening the next phase of the trial in approx. 2 months
  Successful manufacturing of products will be defined initially as the award of a Manufacturers Specials Licence to the CCTL to allow the manufacture of Bone Marrow-Mesenchymal Stromal Cells for compassionate use.
Production of cell-based products to be administered to COVID-19 patients with severe pneumonitis. | Successfully opening the next phase of the trial in approx. 2 months
  Successful manufacturing of products will be subsequently defined by production under MA(IMP) licence, allowing for future production under CTIMP and CTA.
Analysis of cells for understanding production, manufacture and related research. | Successfully opening the next phase of the trial in approx. 2 months
  Successful manufacturing of products, under MA(IMP) licence will be defined as the availability of Bone Marrow-Mesenchymal Stromal Cells to be used in the context of the COMET20 clinical trial.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew McCaskie, FRCS, Principal Investigator — University of Cambridge & Cambridge University Hospitals NHS Foundation Trust
Locations (1):
- Cambridge University Hospitals NHS Foundation Trust, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided